CLINICAL TRIAL: NCT00695734
Title: Interferon-Gamma Release Assays (IGRA) Versus Tuberculin Skin Testing for Detection of Latent Tuberculosis Infection (TB) in Chronic Hemodialysis Patients
Brief Title: Detection of Latent Tuberculosis in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Ligue Pulmonaire Genevoise (Other)
Responsible Party: Jean-Paul Janssens, MD, Division of Pulmonary Diseases; Geneva University Hospital
Other Study IDs: JJanssens 4
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Chronic Renal Failure
Keywords: hemodialysis; end stage renal failure; tuberculosis; latent tuberculosis infection; Patients under hemodialysis for end stage renal failure
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemodialysis: Patients under chronic hemodialysis for chronic end stage renal failure

SUMMARY:
This study aims to compare the performance of the tuberculin skin test, used for more than 50 years as a diagnostic tool for latent tuberculosis infection, with 2 blood tests which have recently become commercially available (Interferon-gamma release assays) in a population of immunosuppressed individuals with chronic renal failure undergoing long term hemodialysis

DETAILED DESCRIPTION:
This prospective study includes all adults aged over 18 years of age who accept to be included in the study and provided written informed consent. All patients are under long term hemodialysis for chronic renal failure. They are subjected to a questionnaire including history of contacts with tuberculosis (TB), prior treatment for TB, history of prior tuberculin skin testing, history of BCG vaccination, country of origin, trips or prolonged stays in high incidence areas, smoking history, and medications. All patients will have a chest X-ray, and simultaneous testing with the tuberculin skin test according to the Mantoux technique, and with the T-SPOT. TB and QuantiFERON Gold in tube Interferon-gamma release assays. The study analysis agreement between tests, detection of prior TB and presumptive latent tuberculosis infection, based on these items.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18
* Under hemodialysis for > 3 months
* End stage renal failure

Exclusion Criteria:

* Refusal to participate
* Prior tuberculin skin test > 15 mm or any adverse reaction to tuberculin skin test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged over 18 Under hemodialysis for > 3 months End stage renal failure
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Relative performance of tuberculin skin test and interferon gamma release assays for detecting latent tuberculosis infection | cross-sectionnal

SECONDARY OUTCOMES:
Agreement between tuberculin skin test and interferon gamma release assays as well as agreement between interferon gamma release assays | cross-sectionnal

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Janssens, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Geneva 14, Switzerland